CLINICAL TRIAL: NCT06859515
Title: A Long-term Follow-up Study to Evaluate the Injection of EXG102-031 Ophthalmic Injection in Participants With Wet Age-related Macular Degeneration (wAMD).
Brief Title: A Long-term Follow up Study of EXG102-031 in Participants With wAMD
Status: Recruiting | Type: Observational
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EXG102-031-111-LTFU
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: AAV; wAMD
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, only for observational studies — No intervention, only for observational studies

SUMMARY:
This is a long-term, safety and efficacy follow-up study of patients in the EXG102-031-111 gene therapy clinical trial for wAMD. Patients will complete visits from the parent study, and then into this long-term follow-up study for continuous safety monitoring for up to 5 years.

DETAILED DESCRIPTION:
This study will enroll patients with wet age-related macular degeneration (wAMD) who have previously be treated with EXG102-031 injection, those patients will Voluntary join this long-term follow-up study to be evaluated the long-term safety and efficacy.

The first two years of long-term follow-up will be conducted every 2 months; From 3 years to 5 years after administration,follow-up visits will be conducted every six months.

ELIGIBILITY:
Inclusion Criteria:

1. Previously received treatment with EXG102-031 in the study (EXG102-031-111);
2. Paticipantes are informed consent and willingness to follow protocol procedures.

Exclusion Criteria:

1. Paticipantes are unwilling or unable to participate in long-term follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: wAMD patients who have previously been treated with EXG102-031 injection in the study (EXG102-031-111).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2030-05-15 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
long-term safety：the types, severity, and incidence of serious adverse events (SAEs), adverse events (AEs). | 4 years
  the types, severity, and incidence of serious adverse events (SAEs), adverse events (AEs).

SECONDARY OUTCOMES:
Change from baseline after treatment by EXG102-031：best corrected visual acuity (BCVA) | 4 years
  Use the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart evaluated. The higher values means better outcome.
Change from baseline after treatment by EXG102-031：central retinal thickness (CRT) | 4 years
  evaluated by Spectral Domain Optical Coherence Tomography (SD-OCT). The higher values means worse outcome.
The times of receiving anti-vascular endothelial growth factor (VEGF) therapy after EXG102-031 administrated | 4 years
  The more times means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei ZHAO, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No